CLINICAL TRIAL: NCT04863391
Title: Pivotal Trial of an Automated AI-based System for Early Diagnosis and Prediction of Late Age Related Macular Degeneration in Primary Care Settings.
Brief Title: Telemedicine in Age-Related Macular Degeneration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The New York Eye & Ear Infirmary (Other)
Collaborators: iHealthScreen Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 18-00787
Record Dates: First submitted 2021-04-19; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- early/none vs.: For identification of early/none (i.e., non-referral level) Age Related Macular Degeneration (ARMD)
  Interventions: Diagnostic Test: Referrable versus Non Referral AMD diagnostic test
- intermediate/late AMD: intermediate/late (i.e., referral level) Age Related Macular Degeneration (ARMD)
  Interventions: Diagnostic Test: Referrable versus Non Referral AMD diagnostic test

INTERVENTIONS:
Diagnostic Test: Referrable versus Non Referral AMD diagnostic test — Artificial intelligence read reports Referrable versus Non Referral AMD

SUMMARY:
This study seeks to evaluate a system for the automated early detection of Age-Related Macular Degeneration (AMD). AMD is a condition in which there is breakdown of the macula of the eye, the part of the retina that is responsible for sharp, central vision. We will take pictures of subjects' eyes using an automated camera. These photographs will be securely transmitted and and then analyzed by a computer program which has been developed in other studies. The outcome of the computer program analysis will be compared with human analysis of these same pictures. If the computer analysis is has good enough accuracy, then this computer system could be used for wide-scale screening for AMD.

DETAILED DESCRIPTION:
iPredict,an AI and telemedicine based software which used individual's color fundus image for early diagnosis of AMD and predict if an individual is at risk of progression to late AMD. iPredict platform integrates the server-side programs (the image analysis and deep-learning modules for AMD severity screening and prediction) and local remote computer/mobile devices (for collecting patient data and images). DRS plus camera will be used in the doctor's office. The remote devices will upload images and data to the server to analyze and screen AMD automatically. The telemedicine platform has been developed for web-based platform. The automatic analysis will be performed on the server, and a report will be sent to the patient/remote devices with an individual's AMD stage as referable or non-referable AMD, and a risk prediction score of developing late AMD (within a minute), and further recommendations to visit a nearby ophthalmologist.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be recruited if willing and able to comply with clinic visit and study-related procedures, and provide signed informed consent
2. Gender of Subjects: Both males and females will be invited to participate.
3. Age of Subjects: Patients will be over 50 years and older

Exclusion Criteria:

1. Unable to provide informed consent.
2. Other retinal degenerations and retinal vascular diseases such as diabetic retinopathy or macular edema, prior retinal surgery.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who fit the eligibility inclusion criteria and not the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-07-19 (Actual); Primary Completion 2022-07-19 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of identification of referable and non-referable AMD for early diagnosis of AMD | 2 years
  Sensitivity of identification of referable and non-referable AMD for early diagnosis of AMD using the iPredict's AI-based AMD screening software utilizing color fundus imaging.
Specificity of identification of referable and non-referable AMD for early diagnosis of AMD using the iPredict's AI-based AMD screening software utilizing color fundus imaging. | 2 years
  Using the gold standard (i.e., the ophthalmologist's grading), the sensitivity and specificity are calculated as: Sens=TP/(TP+FN) Spec=TN/(TN+FP) Where TP is the number of true positives (referable AMD subjects correctly classified), FN is the number of false negatives (referable AMD subjects incorrectly classified as non-referable), TN is the number of true negatives (non-referable subjects correctly classified), and FP is the number of false positives (non-referable AMD subjects incorrectly classified as referable AMD).

CONTACTS AND LOCATIONS:
Locations (1):
- New York Eye and Ear Infirmary of Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no IPD sharing plan at this time.